CLINICAL TRIAL: NCT02575937
Title: The Efficiency of Nutrition Education-based Low Glycemic Diet Intervention on Community Diabetic Patients
Brief Title: Low Glycemic Diet Intervention and Community Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Di Li, Doctor of Medicine, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZXYZM3
Record Dates: First submitted 2015-09-28; First posted 2015-10-15 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes
Keywords: low glycemic diet; diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diabetes group (Experimental): During the trial period, the participants who are diagnosed of diabetes are instructed to consume low glycemic diet every day
  Interventions: Behavioral: low glycemic diet
- Fatty group (Experimental): During the trial period, the participants who are diagnosed of obesity are instructed to consume low glycemic diet every day
  Interventions: Behavioral: low glycemic diet
- Impaired glucose tolerance group (Experimental): During the trial period, the participants who are diagnosed of impaired glucose tolerance are instructed to consume low glycemic diet every day
  Interventions: Behavioral: low glycemic diet

INTERVENTIONS:
Behavioral: low glycemic diet — nutrition education-based low glycemic diet intervention

SUMMARY:
The purpose of this study is to investigate the efficiency of nutrition education-based low glycemic diet intervention on community diabetic patients.

Design: Randomized clinical trial.

Main measures: HbA1c,fasting blood glucose(FBG),2 hours postprandial blood glucose（2hPG）

DETAILED DESCRIPTION:
Low glycemic diet can help to control Blood glucose levels，this study is to investigate the efficiency of nutrition education-based low glycemic diet intervention on community diabetic patients,and to improve health outcomes of patients with type 2 diabetes mellitus (T2DM) by influencing disease self-management through lifestyle modification and diet controlling.

ELIGIBILITY:
Inclusion Criteria:

* subject has a fasting blood glucose between 6.1 and 6.9mmol/L or diagnosed of type 2 diabetes
* glycosylated hemoglobin(A1C) between 6 and 11%.
* subject's age≥18 years.

Exclusion Criteria:

* subject has kidney disease (defined as creatinine>1.3 mg/dl)
* active liver or gallbladder disease
* significant heart disease
* a history of severe hypoglycemia, or use of weight loss medications.
* subject that is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in Glycosylated hemoglobin (HbA1c) | Change from Baseline HbA1c at 12 months
  Because glycosylated hemoglobin is not affected by plasma glucose fluctuation and can reflect the average blood glucose concentration over the past six to eight weeks.We take a blood sample to check participants' glycosylated hemoglobin concentration at baseline and 12 months respectively.Comparing the change of glycosylated hemoglobin levels, to investigate the effect of the our intervention method.

SECONDARY OUTCOMES:
Weight | Baseline and 6, 12 months
Body Mass Index (BMI) | Baseline and 6, 12 months
Fasting blood-glucose | Baseline and 6, 12 months
Total cholesterol level | Baseline and 6, 12 months
HDL level | Baseline and 6, 12 months
LDL level | Baseline and 6, 12 months
Triglycerides | Baseline and 6, 12 months
Food Frequency Questionnaire（FFQ） | Baseline and 6, 12 months
  Method of food frequency questionnaire（FFQ）can be used to monitor the individual over the specified period of time the intake frequencies of certain foods or consumption, so as to determine whether intervention affect their eating habits

CONTACTS AND LOCATIONS:
Overall Officials: Min Xia, PhD, Study Director — Sun Yat-sen University
Locations (1):
- Guangdong Provincial Key Laboratory of Food, Nutrition and Health, Department of Nutrition, School of Public Health, Sun Yat-Sen University (Northern Campus), Guangzhou, Guangdong, China